CLINICAL TRIAL: NCT01683461
Title: Efficacy of HIV Posttest Support for ANC in South Africa
Brief Title: Efficacy of HIV Post-Test Support for ANC in South Africa
Acronym: SAHAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); University of KwaZulu (Other)
Responsible Party: Principal Investigator, Suzanne Maman, Associate Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 07-1070; R01HD050134 (NIH)
Record Dates: First submitted 2012-09-07; First posted 2012-09-11 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: HIV; Acquired Immunodeficiency Syndrome
Keywords: HIV; AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enhanced Counseling (Experimental): Women in the intervention arm receive: (1) a standardized health education video before HIV pre-test counseling; (2) HIV pre- and post-test counseling sessions that prepare women for decisions related to testing, serostatus disclosure and anti-retroviral (ARV) prophylaxis and help women plan strategies for sexual risk behavior change; (3) two additional post-test counseling sessions postpartum focused on legal education and referral, partner testing, sexual risk behavior change and family planning decisions and; (4) an active referral system to post-test support groups run by a clinically trained staff psychologist and (5) an active referral system to legal services run by a lawyer at the clinic.
  Interventions: Behavioral: Enhanced Counseling
- Standard of Care (Active Comparator): Women in the control arm receive the standard of care in terms of HIV counseling and testing during pregnancy. The standard of care for HIV counseling adheres to guidelines provided by the US Centers for Disease Control and the World Health Organization. Women receive one individual pre-test counseling session immediately before they are tested for HIV, and one individual post-test counseling session the same day that they are tested.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Enhanced Counseling — Women in the enhanced counseling arm receive the following intervention package: a video prior to their HIV pre-test counseling session that prepares them for decisions they will have to make regarding HIV testing and PMTCT participation, a pre-test counseling session and post-test counseling session with their nurse midwife/counselor, and two additional post-test counseling sessions with the same nurse midwife at 6 and 10 weeks postpartum. Women in the enhanced counseling arm also have access to ongoing support groups and legal support if needed at the clinic.
  Arms: Enhanced Counseling
Behavioral: Standard of Care — Women in the standard of care arm receive HIV pre and post-test counseling at their first antenatal visit. The counseling provided to them adheres to international guidelines for HIV counseling and testing developed by US CDC and the World Health Organization.
  Arms: Standard of Care

SUMMARY:
This is a randomized controlled intervention trial with 1,500 pregnant and postpartum women to examine the efficacy of an enhanced model of ongoing post-test support for women attending antenatal and postnatal care in KwaZulu-Natal, South Africa. Through the intervention, the investigators will tailor voluntary counseling and testing (VCT) for HIV to the ANC setting and provide a continuum of psychosocial support for pregnant women through: (1) a standardized health education video before HIV pre-test counseling; (2) HIV pre- and post-test counseling sessions that prepare women for decisions related to testing, serostatus disclosure and anti-retroviral (ARV) prophylaxis and help women plan strategies for sexual risk behavior change; (3) two additional post-test counseling sessions postpartum focusing on legal education and referral, partner testing, sexual risk behavior change and family planning decisions and; (4) an active referral system to post-test support groups run by a clinically trained staff psychologist and (5) an active referral system to legal services run by a lawyer at the clinic.

Through this intervention trial the investigators will be testing the following hypotheses:

H1: Women receiving the intervention will have significantly lower sexual risk of HIV at 14 weeks and 9-months post-partum as compared to women in the control arm. Sexual risk of HIV will be measured by: STI incidence (Trichomonas vaginalis, Neisseria gonorrhea and Chlamydia), consistent condom use, unprotected sex in past 30 days, and unprotected sex since delivery.

H2: Women receiving the intervention will report significantly better outcomes related to prevention of mother to child transmission (PMTCT) service uptake at 14 weeks and 9 months post-partum as compared to women in the control arm. PMTCT service uptake will be measured by acceptance of HIV VCT among HIV-positive and HIV-negative women; acceptance of ARVs, adherence to national infant feeding guidelines, and family planning use among HIV-positive women.

H3: Women in the intervention arm will report significantly better psychosocial outcomes at 14 weeks and 9 months post-partum as compared to women in the control arm. Psychosocial outcomes will be measured by: perceived social support, emotional distress, and partner violence among HIV-positive and HIV-negative women.

ELIGIBILITY:
Inclusion Criteria: Eligible women:

1. are at least 18 years old,
2. are not pregnant,
3. have never tested for HIV or had most recently tested negative for HIV at least 3 months prior to recruitment,
4. report having a primary partner who they have been with for at least 6 months,
5. plan to live in Durban for at least the next year,
6. plan to take their infant to the clinic for immunization visits,
7. are able to communicate in English or Zulu, and
8. do not need critical care for a high risk pregnancy that clinic staff is unable to provide.

Exclusion Criteria: Women are ineligible if they:

1. are younger than 18 years;
2. are not pregnant;
3. have previously tested positive for HIV;
4. do not have a primary partner defined as someone they have been with for at least 6 months;
5. are not planning to reside in Durban for the next one year;
6. are unable to communicate in English or Zulu;
7. require care for high risk pregnancy that can not be provided by the clinic staff.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2008-05; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Incidence of sexually transmitted disease | 14 weeks post-partum
  The investigators are using biologic markers of three STIs (Trichomonas vaginalis, Neisseria gonorrhea and Chlamydia). All women are tested for STIs at baseline and 14-weeks post-partum.

SECONDARY OUTCOMES:
Condom use | 14 weeks and 9 months post-partum
  The investigators are measuring consistent condom use, unprotected sex in the past 30 days, unprotected sex since delivery (at 9 months post-partum)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Maman, PhD, Principal Investigator — University of North Carolina, Chapel Hill; Dhayendre Moodley, MMedSc, PhD, Principal Investigator — University of KwaZulu
Locations (1):
- University of KwaZulu-Natal, Durban, South Africa

REFERENCES:
- [Derived] Maman S, Moodley D, McNaughton-Reyes HL, Groves AK, Kagee A, Moodley P. Efficacy of enhanced HIV counseling for risk reduction during pregnancy and in the postpartum period: a randomized controlled trial. PLoS One. 2014 May 13;9(5):e97092. doi: 10.1371/journal.pone.0097092. eCollection 2014. PMID 24824050